CLINICAL TRIAL: NCT02945189
Title: Collection of Urine Samples From Non-pregnant Peri and Post-menopausal Women
Brief Title: Urine Sample Collection From Non Pregnant Peri and Post-menopausal Women
Status: Completed | Type: Observational
Sponsor: SPD Development Company Limited (Industry)
Collaborators: Richmond Pharmacology Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: Protocol-0842
Record Dates: First submitted 2016-10-25; First posted 2016-10-26 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Pregnancy
Keywords: Pregnancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine samples collected and stored
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Peri menopausal: Participants aged 41-55 years
- post menopausal: participants aged 56-65 years

SUMMARY:
This is a sample collection study, participants will be required to collect one (if last menstrual period ≥12 months) or two (if last menstrual period <12 months) urine samples and return them to the study site, together with collection sample information. Participants having a menstrual cycle within the last 6 months will also be required to provide follow-up information on pregnancy status and date of next menstrual bleed.

DETAILED DESCRIPTION:
Each subject will be provided with a urine sample collection container, a transport container, barcode labels, prepaid envelopes and a full set of study instructions, together with the materials required to facilitate the collection of a follow-up urine sample and completion of follow up form, where applicable.

Subjects admitted into the study that are unsure of their pregnancy status will be provided with a marketed Clearblue HPT, to test for pregnancy prior to beginning the study. If a subject informs the trial site that they have become pregnant prior to urine sample collection, they will be withdrawn from the study and no urine sample will be collected. The subject will return their materials to the study site, and the co-ordinator will complete the exit form.

Subjects will be required to collect a urine sample, label their sample (as soon as collected) with the appropriate bar-coded label provided and return this to the study site. Where it is not possible to return the sample as soon as collected, urine samples must be stored in a domestic fridge in the container provided for a maximum of 1 week and then sent to the study site at their earliest convenience.

Subjects will receive follow-up to establish pregnancy status unless ≥ 12 months from their last menstrual period (LMP). On completion of the study, subjects will be reimbursed for their participation.

It is anticipated that sample collection will be carried out remotely (i.e. at the volunteers home) but volunteers may attend the study site for sample collection should they require.

ELIGIBILITY:
Inclusion Criteria:

* Known to be not pregnant,
* Willing to give consent

Exclusion Criteria:

* Pregnant or breastfeeding,
* Pregnant within last 2 months,
* Having treatment for infertility,
* Taken hormonal contraception containing hCG in last month,
* Using hormonal contraception within last month,
* Previously taken part in sample collection study for SDP (providing 1-7 samples).

Ages: 41 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 443 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Individual urine samples obtained from 150 not pregnant women aged 41-55 years and 150 not pregnant women aged 56 - 65 years | 2 months
  Urine sample collection from healthy volunteers of peri (age 41-55) and post (age 56-65) menopausal women

CONTACTS AND LOCATIONS:
Overall Officials: Jorg Taubel, MD FFPM, Principal Investigator — Richmond Pharmacology

IPD SHARING:
Plan to Share IPD: No
This is a sample collection study only, no research IPD available